CLINICAL TRIAL: NCT00655967
Title: Safety of Acamprosate for Alcohol Dependence in the Elderly: An Open-Label Study
Brief Title: Safety of Acamprosate for Alcohol Dependence in the Elderly: An Open-Label Study (SAFADIE)
Acronym: SAFADIE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRRC# 06-318; CMP-MD-11
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Acamprosate(Campral)
  Interventions: Drug: Acamprosate (Campral); Drug: Acamprosate

INTERVENTIONS:
Drug: Acamprosate (Campral) — During the course of the study patients will be supplied with 333mg tablets of acamprosate provided by the Sponsor. The study medication will be administered at a dose of 666mg (=two tablets) three times a day for patients with a creatinine clearance >50. The dose will be 333mg three times a day for patients with a creatinine clearance in the range of 30-50.
  Treatment compliance will be monitored by counts of returned medication. Records of all concomitant medications will be taken at each study visit as well as reports of adverse events (as shown above).
  Other Names: Acamprosate(Campral)
Drug: Acamprosate — During the course of the study patients will be supplied with 333mg tablets of acamprosate provided by the Sponsor. The study medication will be administered at a dose of 666mg (=two tablets) three times a day for patients with a creatinine clearance >50. The dose will be 333mg three times a day for patients with a creatinine clearance in the range of 30-50.
  Other Names: Acamprosate(Campral)

SUMMARY:
Alcohol abuse and dependence are very prevalent and result in significant morbidity, mortality and cost to society (Harwood 2000). Pharmacotherapies to assist with alcohol dependence consist of disulfiram, naltrexone and acamprosate. Of these, acamprosate is unique in that it is not metabolized by the liver, but rather completely excreted renally. In contrast, naltrexone is metabolized by the CYP450 system of the liver and less than 2% is excreted unchanged and can cause liver damage (PDR 2005). Multiple cases of hepatitis, including both cholestatic and fulminant hepatitis, as well as hepatic failure resulting in transplantation or death, have been reported with administration of disulfiram (PDR 2005). The incidence of liver disease among alcoholics is high and increases with age and years of drinking and this may preclude the use of antabuse or naltrexone to help alcohol dependent patients with liver disease or that are elderly . Thus acamprosate has a unique safety profile that would make it ideally suited for treating alcohol dependence in the elderly, even in the presence of hepatic impairment. The current study is to evaluate the safety profile of acamprosate in elderly patients with alcohol dependence.

Acamprosate, calcium acetyl homotaurinate, has been approved in most European countries and the U.S. for the maintenance of abstinence in recently detoxified alcoholics. The mechanism of action involves primarily the restoration of a normal N-methyl- D -aspartate (NMDA) receptor tone in glutamatergic systems (Rammes et al 2001). Several trials of acamprosate confirm its efficacy in the maintenance of abstinence in alcohol dependence (Lesch et al. 2001; Slattery et al. 2003; Mann et al. 2004; Verheul et al. 2004). It also reduces the severity of relapse in alcoholics in abstinence based treatment programs (Chick et al. 2003). There is limited data on the safety of acamprosate in the elderly (PDR 2005).

For the purposes of this study, elderly will be defined as 60 years or older.

STUDY OBJECTIVE: To determine the short-term safety of Acamprosate in the treatment of alcohol dependence in the elderly.

DETAILED DESCRIPTION:
STUDY DESIGN: This trial will be conducted as an open-label, fixed dose design for safety of Acamprosate in the elderly. Subjects will receive Acamprosate for 12 weeks. The schedule of visits will include screening, baseline and three monthly follow-up visits at days 30, 60 and 90. We will recruit 25 subjects in the total study period of 15 month.

Regarding the number of subjects, chi-squared analysis of the total number of side effects (61%, i.e. 1230 out of 2018 subjects in prior studies) and the possible number of subjects in the study with side effects (from 0 to 25), indicates that a significant (alpha=0.05) difference from the previously observed rate would occur if less than 11 (p<=0.05) or more than 20 (p<=0.025) subjects report side effects. Side effects in 11 to 20 subjects would be nonsignificantly different from the previously published rates. Thus 25 subjects are sufficient to detect significant deviation in frequency of overall side effects in this sample compared to the subjects in prior studies. Total number of side effects was used for this calculation because there is no single common or significant side effect that would lend itself as an appropriate surrogate for the side effects overall.

During the course of the study subjects will be supplied with 333mg tablets of Acamprosate provided by the Sponsor. The study medication will be administered at a dose of 666mg (=two tablets) three times a day for subjects with a creatinine clearance >50. The dose will be 333mg three times a day for subjects with a creatinine clearance in the range of 30-50.

Safety will be monitored by subject's report of adverse events at all treatment visits throughout both, open label and double blind phases of the Trial. The report of adverse events or new symptoms by the subject will be reviewed and summarized. This may also include any clinically significant changes in the vital signs (blood pressure and pulse readings, weight, temperature), physical examinations, laboratory evaluations (blood chemistry, hematology, urinalysis, EKG) and recording of concomitant treatment. A DSMB plan has been set up.

Treatment compliance will be monitored by counts of returned medication, and subjects are to be counseled if they do not adhere, or if they are thought to be at risk for not adhering to the medication regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, men and women, age 60 and older.
2. Patients with Alcohol Dependence as determined by SCID I section for substance use disorders who are not in full sustained remission.
3. Patients who have consumed significant amounts of alcohol in the past 30 days, as determined by Time Line Follow Back report by patient and patient's spouse, partner or friend. Significant amounts is defined for these purposes as at least one episode of 5 or more drinks, with a drink defined as one bottle of beer, one glass of wine or one shot of liquor.
4. Patients, who are able to comprehend and satisfactorily comply with protocol requirements.
5. Patients, who signed the written informed consent given prior to entering any study procedure and completed the informed consent quiz.

Exclusion Criteria:

1. Patients with the following concurrent DSM-IV Axis I diagnoses as determined by the relevant sections of SCID I:

   * Current, acute psychosis regardless of etiology
   * Moderate to severe dementia regardless of etiology, defined as a MMSE score of 18 or less out of 30.
   * Current opioid, cocaine or amphetamine dependence, defined as not meeting criteria for sustained full remission.
2. Patients with significant or unstable medical conditions as determined by investigator. This is defined as a medical condition that, in the Investigator's opinion, would expose them to an increased risk of a significant adverse event or interfere with assessments of safety during the course of the trial.
3. Patients with significantly abnormal lab values, as determined by the investigator, including creatinine clearance less than 30 as determined by Cockcroft-Gault estimate.
4. Patients with a history of intolerance or hypersensitivity to acamprosate.
5. Patients who are actively suicidal.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be safety. | Patients will receive acamprosate for 12 weeks.The schedule of visits will include screening, baseline and and three monthly follow-up visits at days 30, 60 and 90. We will recruit 25 subjects in the total study period of 12 month.

SECONDARY OUTCOMES:
Changes in the quantity of alcohol consumed as determined by Time Line Follow Back assessment by patient and parallel historian will be determined. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Florian Birkmayer, M.D., Principal Investigator — University of New Mexico, Department of Psychiatry
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States